CLINICAL TRIAL: NCT00221884
Title: Does Ultrasound Guidance Improve the Success of Brachial Plexus Block? A Prospective, Randomized, Controlled Trial.
Brief Title: Use of Ultrasound in Upper Extremity Blocks.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Anesthesiologists' Society (Other); The Physicians' Services Incorporated Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UHN02-0430-E
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2005-09

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — High-Energy Shock Waves

INTERVENTIONS:
Procedure: Ultrasound

SUMMARY:
Many patients undergoing surgery on their hand receive a form of anesthetic called "axillary brachial plexus block". This involves the injection of local anesthetic (freezing medication) around the nerves that supply the upper limb, which are located in the arm pit. The technique currently used by physicians performing this procedure is far from perfect, and in up to 1 of every 5 patients it does not work well enough to allow surgery, and a different form of anesthetic may need to be used.

In an attempt to improve these results, we have recently developed a new technique, using ultrasound imaging to "see" the nerves prior to giving the injection. Our initial results are very promising, implying that this may be a highly successful and safe approach. The purpose of this study is to determine if this technique is indeed more successful. In order to do that, we will ask 110 patients for their participation. They will be divided in two groups, at random. One group will receive the standard technique (transarterial, using a small needle to find the artery that is close to the nerves). The other group will receive the injection after identifying the nerves with ultrasound imaging. They will all receive the same type of medication, and they will be tested every 5 minutes for half an hour to determine if the block has been successful, according to pre-established criteria. Their pain control will be assessed after the surgery and they will be called 24 hours and 1 week after the surgery to assess their recovery and rule out any possible complications.

DETAILED DESCRIPTION:
Ultrasonography has been used successfully to define the anatomy of the brachial plexus in the interscalene, supraclavicular and axillary regions. This is a widely available technology, it is non-invasive, portable, less expensive than other imaging modalities and allows for real time imaging simultaneously with the block procedure.

There are some recent case reports and small case series describing the use of ultrasound to image the brachial plexus and to guide brachial plexus blockade 16,17,18. We have used ultrasound imaging to succesfully identify the brachial plexus and guide needle localization and nerve stimulation in 15 volunteers 19. In these healthy volunteers, we were able to identify the brachial plexus in every subject, at four different anatomical levels : interscalene, supraclavicular, axillary and mid-humeral (see figures). Needle localization and nerve stimulation were also successful in every case. Moreover, preliminary data from an ongoing series at our institution, shows that when ultrasound guidance is used, supraclavicular brachial plexus block can be performed with a high success rate (97%)20.

However, whether ultrasound guidance truly improves success rates when compared to more traditional techniques is still unknown. There has been no randomized controlled trial published to date addressing this question.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3
* 18 to 80 years of age
* 50 to 100 kg of body weight
* elective upper extremity procedure amenable to brachial plexus block
* estimated surgical time > 1 hr

Exclusion criteria

* Any medical contraindication to brachial plexus block ( allergy to local anesthetics, coagulopathy, loco-regional malignancy or infection, neurological deficit in the area to be blocked, severe respiratory disease)
* Inability to read, write or speak English
* Chronic pain longer than 6 months
* Chronic opioid use
* History of drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-08; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent WS Chan, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada